CLINICAL TRIAL: NCT02285010
Title: Effects of Pre-operative Oral Pregabalin on Post Operative Morphine Consumption After Abdominal Hysterectomy With/Without Salpingo-oophorectomy Under Spinal Anesthesia With Intrathecal Morphine
Brief Title: Effect of Pregabalin on Post Operative Pain in Abdominal Hysterectomy Under Spinal Anesthesia With Intrathecal Morphine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Si594/2014
Record Dates: First submitted 2014-10-31; First posted 2014-11-06 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Post Operative Pain
Keywords: pregabalin; postoperative pain; abdominal hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo in capsule is prescribed to the patient 60 min prior to the surgery.
  Interventions: Drug: placebo
- Pregabalin (Active Comparator): Pregabalin (150 mg) one capsule is prescribed to the patient 60 min prior to the surgery.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: placebo — Placebo in capsule is prescribed to the patient 60 min prior to the surgery. Ringer Lactate Solution preload 15 mL/kg prior to surgery. Spinal anesthesia is done with 0.5% Heavy bupivacaine + morphine 0.2 mg total volume 3.0 - 3.6 mL. IV PCA Morphine is applied at PACU (bolus dose only 1 mg, lockout interval 5 min, 4 hr limit 35 mg). As soon as the patient is allowed to sip, paracetamol (500 mg) 1 tab PO every 6 hours is prescribed.
  Arms: Placebo
Drug: Pregabalin — Pregabalin (150 mg) one capsule is prescribed to the patient 60 min prior to the surgery.
  Ringer Lactate Solution preload 15 mL/kg prior to surgery. Spinal anesthesia is done with 0.5% Heavy bupivacaine + morphine 0.2 mg total volume 3.0 - 3.6 mL. IV PCA Morphine is applied at PACU (bolus dose only 1 mg, lockout interval 5 min, 4 hr limit 35 mg). As soon as the patient is allowed to sip, paracetamol (500 mg) 1 tab PO every 6 hours is prescribed.
  Other Names: Lyrica
  Arms: Pregabalin

SUMMARY:
This study aims to compare the effect of pre-operative oral pregabalin on post operative morphine consumption after abdominal hysterectomy with/without salpingo-oophorectomy.

DETAILED DESCRIPTION:
The participants are randomized into two groups by computer randomization. The patient undergo spinal anesthesia with 0.5% Heavy bupivacaine with morphine 0.2 mg. IV PCA morphine is initiate in the post-anesthetic care unit. We compare post operative morphine consumption in the first 24 hours, time to first analgesia, adverse event, and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

1. ASA classification 1-2 undergoing abdominal hysterectomy with/without salpingo-oophorectomy under spinal anesthesia with intrathecal morphine
2. Patient can use patient-controlled analgesia (IV PCA)

Exclusion Criteria:

1. History of drug allergy to gabapentinoid and related drug
2. History of regular analgesic drug use, psychiatric drug usage, drug abuse, alcohol addiction or chronic pain patient
3. Renal disease (Creatinine Clearance < 60), Liver disease, Seizure disorder and Psychiatric disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taniga Kiatchai, MD, Principal Investigator — Mahidol University
Locations (1):
- Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Background] Schmidt PC, Ruchelli G, Mackey SC, Carroll IR. Perioperative gabapentinoids: choice of agent, dose, timing, and effects on chronic postsurgical pain. Anesthesiology. 2013 Nov;119(5):1215-21. doi: 10.1097/ALN.0b013e3182a9a896. No abstract available. PMID 24051389
- [Background] Sahgal N, Banerjee A. Efficacy of pregabalin in acute postoperative pain: a meta-analysis. Br J Anaesth. 2011 Aug;107(2):274; author reply 275. doi: 10.1093/bja/aer207. No abstract available. PMID 21757554
- [Background] Engelman E, Cateloy F. Efficacy and safety of perioperative pregabalin for post-operative pain: a meta-analysis of randomized-controlled trials. Acta Anaesthesiol Scand. 2011 Sep;55(8):927-43. doi: 10.1111/j.1399-6576.2011.02471.x. Epub 2011 Jun 27. PMID 21707548

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 142 patients on gynecology unit during December 2014 - January 2016 were assessed for eligibility, 17 patient were not randomized due to didn't meet inclusion criteria (n=6), met exclusion criteria (n=4), declined to participate (n=7).
Groups:
- Placebo: Placebo in capsule is prescribed to the patient 60 min prior to the surgery.
  placebo: Placebo in capsule is prescribed to the patient 60 min prior to the surgery.
  Ringer Lactate Solution preload 15 mL/kg prior to surgery. Spinal anesthesia is done with 0.5% Heavy bupivacaine + morphine 0.2 mg total volume 3.0 - 3.6 mL. IV PCA Morphine is applied at PACU (bolus dose only 1 mg, lockout interval 5 min, 4 hr limit 35 mg). As soon as the patient is allowed to sip, paracetamol (500 mg) 1 tab PO every 6 hours is prescribed.
- Pregabalin: Pregabalin (150 mg) one capsule is prescribed to the patient 60 min prior to the surgery.
  Pregabalin: Pregabalin (150 mg) one capsule is prescribed to the patient 60 min prior to the surgery.
  Ringer Lactate Solution preload 15 mL/kg prior to surgery. Spinal anesthesia is done with 0.5% Heavy bupivacaine + morphine 0.2 mg total volume 3.0 - 3.6 mL. IV PCA Morphine is applied at PACU (bolus dose only 1 mg, lockout interval 5 min, 4 hr limit 35 mg). As soon as the patient is allowed to sip, paracetamol (500 mg) 1 tab PO every 6 hours is prescribed.
Period: Overall Study
Arm/Group | Placebo | Pregabalin
Started | 63 | 62
Completed | 58 | 61
Not Completed | 5 | 1
Not completed — not abdominal hysterectomy | 2 | 0
Not completed — Not spinal anesthesia | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin | Total
Number analyzed (Participants) | 58 | 61 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (6.1) | 45.9 (5.3) | 46.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 61 | 119
  Male | 0 | 0 | 0
ASA physical status [Count of Participants; unit: Participants] — ASA American Society of Anesthesiologists; ASA I - Healthy patient, ASA II - Patient with controlled systemic disease (higher ASA status means more complicated patient)
  Participants
    I | 35 | 27 | 62
    II | 23 | 34 | 57

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Morphine Consumption
Description: Cumulative morphine consumption in the first 24 hours is recorded from IV PCA
Time Frame: 6, 12, and 24 hours after operation
Population: Only 47 and 53 participants from placebo and pregabalin group, respectively, received IV-PCA morphine in the 1st 24 hours. The rest didn't require morphine consumption.
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 47 | 53
mg
  Morphine consumption 6 hr | 1 [0 to 3.3] | 0 [0 to 2]
  Morphine consumption 12 hr | 1 [0 to 4] | 1 [0 to 4.5]
  Morphine consumption 24 hr | 4 [1.8 to 10] | 5 [2 to 11]
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Non-Inferiority — Definition: 50% reduction of morphine consumption Type I error (alpha) 0.05, Type II error (beta) 80%; p = 0.60, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Time to First Analgesia
Description: Time to first analgesia is recorded from IV PCA.
Time Frame: 24 hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 47 | 53
hour | 4.6 [2.1 to 23.9] | 7.7 [2.5 to 23.7]
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Non-Inferiority — Alpha 0.05, Beta 80%; p = 0.10, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Pain Scores on the Visual Analog Scale
Description: Pain score is evaluated by nurses using Numerical Rating Scale (NRS)
  Minimum score 0 (no pain), Maximum score 10 (worst imaginable pain), lower scores mean a better outcome
Time Frame: 24 hours
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 58 | 61
score on a scale
  At rest | 2 [0 to 4] | 2 [0 to 3]
  At movement | 4 [2 to 6] | 4 [3 to 5]
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; for NRS at rest; Test type: Non-Inferiority — alpha 0.05, beta 80%; p = 0.33, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; for NRS at movement; Test type: Non-Inferiority — alpha 0.05, beta 80%; p = 0.75, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Numbers of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Measure sedation score by evaluate and observe; measure pruritus, PONV, dizziness, visual disturbance using questionnaire
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 58 | 61
Participants
  Pruritus: No | 7 | 17
  Pruritus: Mild | 35 | 31
  Pruritus: Moderate | 15 | 10
  Pruritus: Severe | 1 | 3
  Nausea: No | 18 | 23
  Nausea: Mild | 24 | 21
  Nausea: Moderate | 16 | 17
  Nausea: Severe | 0 | 0
  Vomiting: No | 31 | 38
  Vomiting: Mild | 10 | 9
  Vomiting: Moderate | 12 | 8
  Vomiting: Severe | 5 | 6
  Dizziness: No | 18 | 14
  Dizziness: Mild | 31 | 39
  Dizziness: Moderate | 9 | 7
  Dizziness: Severe | 0 | 1
  Visual disturbance: No | 51 | 45
  Visual disturbance: Mild | 7 | 16
  Visual disturbance: Moderate | 0 | 0
  Visual disturbance: Severe | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; For pruritus; Test type: Non-Inferiority — alpha 0.05, beta 80%; p = 0.16, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; For Nausea; Test type: Non-Inferiority — Alpha 0.05, beta 80%; p = 0.66, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs Pregabalin; For Vomiting; Test type: Non-Inferiority — alpha 0.05, beta 80%; p = 0.46, Chi-squared
Statistical Analysis 4: Comparison: Placebo vs Pregabalin; For Dizziness; Test type: Non-Inferiority — Alpha 0.05, beta 80%; p = 0.54, Chi-squared
Statistical Analysis 5: Comparison: Placebo vs Pregabalin; For visual disturbance; Test type: Non-Inferiority — Alpha 0.05, beta 80%; p = 0.05, Chi-squared

5. Secondary Outcome: Number of Patients Evaluating Their Satisfaction
Description: Using four-point scale to evaluate patient satisfaction. Patients indicated if their satisfaction was Unsatisfied, Less Satisfied, Moderately Satisfied, or Good Satisfied.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 58 | 61
Participants
  Unsatisfied | 0 | 0
  Less satisfied | 1 | 5
  Moderate satisfied | 19 | 25
  Good satisfied | 38 | 31
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Non-Inferiority — Alpha 0.05, beta 80%; p = 0.05, Chi-squared — P-Value 0.05 was calculated

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | Placebo | Pregabalin
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/62
Other Adverse Events (participants affected / at risk) | 0/63 | 0/62

LIMITATIONS AND CAVEATS:
1. Did not perform intention-to-treat analysis. When the treatment plan was changed, the patient was withdrawn from the study.
2. Single dose pre-operation instead of multi-dose post-operation.
3. Homogeneity of population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes